CLINICAL TRIAL: NCT03722771
Title: Influence of Lavender Oil on Vital Signs and Anxiety in Oral Surgery Patients: a Randomized Controlled Clinical Trial
Brief Title: Influence of Lavender Oil on Vital Signs in Oral Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazife Begüm KARAN (Other)
Responsible Party: Sponsor-Investigator, Nazife Begüm KARAN, Assistant Professor, DDS, PhD, Recep Tayyip Erdogan University Training and Research Hospital
Organization: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 106
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Dental Anxiety; Sedative; Anxiety Disorder
Keywords: Lavandula; phytotherapy; aromatherapy; dental anxiety; anaesthesia
MeSH Terms: conditions — Anxiety Disorders | interventions — Inhalation; Blood Pressure; Respiratory Rate; Heart Rate; Oxygen Saturation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lavender oil group (A) (Experimental): 100 % pure, high strength lavender oil inhalation in a separate room for 3 minutes, prior to surgery.
  Anxiety questionnaires 1 (MDAS) Anxiety questionnaires 2 (STAI-S) Vital signs 1 (Blood pressure) Vital signs 2 (respiratory rate,) Vital signs 3 (heart rate) Vital signs 4 (saturation)
  Interventions: Behavioral: Inhalation; Other: Anxiety Questionnaires 1; Other: Anxiety Questionnaires 2; Diagnostic Test: Vital Signs 1; Diagnostic Test: Vital Signs 2; Diagnostic Test: Vital Signs 3; Diagnostic Test: Vital Signs 4
- control group (B) (Sham Comparator): No application of lavender oil, prior to surgery. Anxiety questionnaires 1 (MDAS) Anxiety questionnaires 2 (STAI-S) Vital signs 1 (Blood pressure) Vital signs 2 (respiratory rate,) Vital signs 3 (heart rate) Vital signs 4 (saturation)
  Interventions: Other: Anxiety Questionnaires 1; Other: Anxiety Questionnaires 2; Diagnostic Test: Vital Signs 1; Diagnostic Test: Vital Signs 2; Diagnostic Test: Vital Signs 3; Diagnostic Test: Vital Signs 4

INTERVENTIONS:
Behavioral: Inhalation — lavender oil inhalation in a separate room for 3 minutes prior to surgery
  Other Names: lavender oil application
  Arms: lavender oil group (A)
Other: Anxiety Questionnaires 1 — Modified Dental Anxiety Scale was used to describe the level of the dental anxiety.
  Other Names: Modified Dental Anxiety Scale
Other: Anxiety Questionnaires 2 — State-Trait Anxiety Inventory-State Scale was used to distinguish the true anxiety level of the patients from the anxiety level for a particular situation.
  Other Names: State-Trait Anxiety Inventory-State Scale
Diagnostic Test: Vital Signs 1 — Changes in vital signs 1 - blood pressure - before, during and after the procedure were noted.
  Other Names: Blood Pressure
Diagnostic Test: Vital Signs 2 — Changes in vital signs 2 - respiratory rate - before, during and after the procedure were noted.
  Other Names: Respiratory rate
Diagnostic Test: Vital Signs 3 — Changes in vital signs 3 - heart rate - before, during and after the procedure were noted.
  Other Names: Heart rate
Diagnostic Test: Vital Signs 4 — Changes in vital signs 4 - saturation - before, during and after the procedure were noted.
  Other Names: Saturation

SUMMARY:
The aim of this study is to investigate the impact of lavender oil (Lavandula angustifolia) on anxiety, mood, vital signs (blood pressure, respiratory rate, heart rate and saturation) for oral surgery patients.

DETAILED DESCRIPTION:
Lavender oil has sedative properties. Oral surgical procedures have been proven as to be the greatest concern among dental practices for patients. Limited randomized clinical trials have demonstrated evidence-based results of lavender oil, despite being the most effective essential oil for anxiety and stress. The hypothesis of the present study was that the inhalation of lavender oil prior to oral surgical procedures may reduce anxiety and consequently may effect intra and post-operative blood pressure, inspiration and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of wisdom tooth
* Must be similar in age-height-weight
* Must be similar socio-culturally

Exclusion Criteria:

* Under 18 years of age
* Taking psychotropic medication or psychiatric treatment
* Systemically unhealthy patients
* Pregnants

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Vital Sign Measurements - 1 - changes in blood pressure | through study completion an average of 3 months
  changes in blood pressure
Vital Sign Measurements - 2 - changes in respiratory rate | through study completion an average of 3 months
  changes in respiratory rate
Vital Sign Measurements - 3 - changes in heart rate | through study completion an average of 3 months
  changes in heart rate
Vital Sign Measurements - 4 - changes in saturation level | through study completion an average of 3 months
  changes in saturation level

SECONDARY OUTCOMES:
Anxiety Test 1 - MDAS tests | through study completion an average of 3 months
  MDAS tests
Anxiety Test 2 - STAI-S tests | through study completion an average of 3 months
  STAI-S tests

CONTACTS AND LOCATIONS:
Overall Officials: Nazife Begüm KARAN, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Nazife Begüm KARAN, Rize, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karan NB. Influence of lavender oil inhalation on vital signs and anxiety: A randomized clinical trial. Physiol Behav. 2019 Nov 1;211:112676. doi: 10.1016/j.physbeh.2019.112676. Epub 2019 Sep 7. PMID 31505191